CLINICAL TRIAL: NCT05621330
Title: Efficacy and Safety of QL0911 in Adult Patients With Chronic Primary Immune Thrombocytopenia: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase III Trial
Brief Title: Efficacy and Safety of QL0911 in Adult Patients With Chronic Primary Immune Thrombocytopenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QL0911-003
Record Dates: First submitted 2022-11-10; First posted 2022-11-18 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Primary Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL0911 (Experimental)
  Interventions: Drug: QL0911
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: QL0911 — The study in a 2:1 randomization ratio(144 subjects to QL0911). Qilu investigational product (QL0911 or placebo) will be administered in the clinic by a qualified healthcare provider as a subcutaneous injection.
  Arms: QL0911
Drug: Placebo comparator — The study in a 2:1 randomization ratio(72 subjects to Placebo ). Qilu investigational product (QL0911 or placebo) will be administered in the clinic by a qualified healthcare provider as a subcutaneous injection.
  Arms: Placebo

SUMMARY:
QL0911, a recombinant human thrombopoietin mimetic peptide-Fc fusion protein for injection, is a romiplostim (Nplate®) biosimilar for the treatment of primary immune thrombocytopenia (ITP). This phase III study aimed to assess the efficacy and safety of QL0911 in adult patients with primary chronic ITP.

DETAILED DESCRIPTION:
This study consisted of a randomized, double-blind, placebo-controlled, 26-week treatment period, sequentially followed by an open-label, single-arm, 12-week treatment period, and an additional 4-week safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years old;
* Diagnosed primary ITP for at least 12 months;
* Had received at least one first-line ITP treatment with no response or recurrence after treatment;
* Had a platelet count <30×10^9/L within 48 hours before the first dose;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2;
* Fully understand and comply with the requirements of this study, and voluntarily sign the informed consent form.

Exclusion Criteria:

* Had a history of bone marrow stem cell abnormalities or myelodysplastic syndrome other than ITP-specific changes.
* Had arterial thrombosis, or venous thromboembolism; severe cardiovascular diseases; malignant tumors; secondary thrombocytopenia caused by autoimmune diseases.
* Underwent splenectomy within 12 weeks before the first dose;
* Had received ITP treatments (including rescue treatment) within 2 weeks before the first dose;
* Had received romiplostim (Nplate®) or eltrombopag (Revolade®), rhTPO or other agents that stimulate TPO receptors (also known as c-Mpl), and hematopoietic growth factors (HGFs) within 4 weeks before the first dose;
* Had received antineoplastic agents within 8 weeks before the first administration, but when treating ITP with hypomethylating agents (HMA) such as decitabine, a 4-week washout period was acceptable, as judged by the investigator;
* Had received antibody-based therapies within 14 weeks before the first dose; 8) had serum creatinine or total bilirubin >1.5 upper limit of normal (ULN), alanine transaminase (ALT) or aspartate transaminase (AST) >3 ULN, hemoglobin < 100g/L, absolute neutrophil count <1.5x10^9/L;
* Had prothrombin time (PT) or prothrombin time-international normalized ratio (PT-INR) or activated partial thromboplastin time (APTT) exceeded 20% of the reference range of normal values.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
proportion of patients achieving durable platelet response at week 24 during the double-blind treatment period | 24weeks

SECONDARY OUTCOMES:
proportion of patients with weekly platelet responses within 24 weeks of treatment; | 24weeks
Proportion of patients who achieved platelet count ≥ 30 × 10^9/L at least a two-fold increase from baseline platelet count without bleeding during the 24-week double-blind period; | 24weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Shandong, China

REFERENCES:
- [Derived] Zhou H, Han S, Jin J, Huang R, Guo X, Shen X, Wang B, Wang X, Yao H, Du X, Huang M, Ran X, Wang W, Yang T, Zhang F, Zheng C, Zuo X, Fu R, Gao D, Ge Z, Han Y, Li Y, Kang X, Shi Y, Hou M. Efficacy and safety of QL0911 in adult patients with chronic primary immune thrombocytopenia: A multicenter, randomized, double-blind, placebo-controlled, phase III trial. J Transl Int Med. 2023 Dec 20;11(4):423-432. doi: 10.2478/jtim-2023-0106. eCollection 2023 Dec. PMID 38130645